CLINICAL TRIAL: NCT02570958
Title: Robotic ICG Guided Surgery (RIGGS) Using Electromagnetic Navigational Bronchoscopy (ENB): A Novel Technique for Targeting Small Lung Tumors
Brief Title: ENB Robotic ICG Guided Surgery: A Novel Technique for Targeting Small Lung Tumors
Acronym: ENB-RIGGS
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Funding was not received
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Principal Investigator, Wael Hanna, Director, Research Program, Boris Family Centre for Robotic Surgery, St. Joseph's Healthcare Hamilton
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BFCRS-RP-002-1504-29
Record Dates: First submitted 2015-10-06; First posted 2015-10-07 (Estimated); Last update posted 2017-06-05 (Actual); Status verified 2017-06

CONDITIONS: Non-small Cell Lung Cancer; Thoracic Surgery
Keywords: robotic surgery; indocyanine green; electromagnetic navigational bronchoscopy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Indocyanine green (Experimental)
  Interventions: Drug: Indocyanine Green

INTERVENTIONS:
Drug: Indocyanine Green — In the operating room ENB will be used to locate the targeted lung tumor. Once the tumor is located, the surgeon will advance a bronchoscope to the tumor, a needle will be passed through the bronchoscope, and the tumor will be injected with 100-150 micro liters of ICG solution at 0.125mg/mL concentration. The tumor is expected to fluoresce using the da Vinci Firefly robotic camera, giving off a bright green hue. Wedge resection of the fluorescent part of the lung will then be performed. The excised specimen will be sent for immediate pathologist analysis. If the tumor is found within the specimen, and the specimen margins are free of tumor cells, then the procedure will be completed. If the tumor cannot be targeted or visualized, or if the tumor is not found in the pathological specimen, or if the margins of the specimen contain tumor cells, then a formal anatomical lobectomy or segmental resection of the lung will be performed to ensure that the tumor is completely excised.
  Other Names: IC-GREEN

SUMMARY:
Lung cancer is the leading cause of cancer deaths worldwide. However, if diagnosed at an early stage (tumor <2 cm), lung cancer is highly curable with a 5-year survival rate greater than 80% after surgical resection. Screening tests have made it easier to identify small lung tumors. However, these tumors are often not visible to the naked eye, and surgeons cannot feel them, making them difficult to precisely locate and remove. For this reason, surgeons have become more reliant on image guided surgery for the removal of these tumors.

The standard of care for locating and removing small lung tumors is microcoil-guided video-assisted thoracoscopic surgery (VATS). This is a two-step procedure performed by two separate physicians.

* First, patient is taken to radiology suite and radiologist inserts a microcoil near the lung tumor
* Second (usually occurs a few hours later), patient is taken to operating room; a surgeon uses an x-ray arm to find the microcoil within the lung and remove it surgically.

A pathologist reviews the resected tissue to make sure that the tumor and the microcoil were both removed. Until this evaluation, the surgeon does not know whether the tumor has been removed or not. While this method is safe, it is time consuming, uses staff resources, and requires bulky equipment to complete.

In this study, we plan to develop and test a new method of identifying and removing small lung tumors. This procedure is called Electromagnetic Navigational Bronchoscopy (ENB) Robotic Indocyanine Green Guided Surgery (RIGGS) or ENB-RIGGS for a short name. The purpose of this study is to test the safety and reliability of the ENB-RIGGS surgery in the form of a pilot study.

ENB-RIGGS surgery is done in the operating room by a surgeon under general anesthetic. ENB-RIGGS begins by creating a 3-D GPS map of the lung which guides the surgeon directly to the tumor. A fluorescent green dye called indocyanine green is then injected into the tumor, and when viewed by the special robotic camera the tumour will fluoresce with a green hue allowing the surgeon to easily see the tumour. The surgeon then uses the robot to remove the tumor and surrounding tissue. The lung tissue specimen will be evaluated immediately by a pathologist.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. Peripheral lung tumour that is <2 cm in size on a CT scan
3. Fit to undergo thoracic surgery as assessed by the surgeon.

Exclusion Criteria:

1. Hypersensitivity or allergy to ICG, sodium iodide or iodine
2. Women who are currently pregnant or are breast feeding; or women of child bearing potential who are not currently taking adequate birth control.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-10 (Estimated); Primary Completion 2017-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Safety determined by the rates of adverse reactions to ICG dye, intra-operative adverse events, and post-operative complications as defined by the Ottawa Thoracic Morbidity and Mortality classification | Post-operatively, an average of 2 years
Reproducibility | Post-operatively, an average of 2 years
  Reproducibility will be measured by the aggregate score on items 1-4 of the 6-item scale which include: targeting of tumor on ENB (advance a bronchoscope to the targeted tumor); injection of the tumour with ICG; detection of ICG fluorescence with near-infrared light; wedge resection. The reproducibility score for each procedure will be the sum of the first 4 items on the 6-item scale and can range between 0/4 to 4/4. The reproducibility rate will be defined as the percentage of patients who score 4/4 on the reproducibility scale.
Oncological validity | Post-operatively, an average of 2 years
  The oncological validity score for each procedure will be the sum of the last 2 items on the 6-item scale (ex-vivo localization of tumor; ex-vivo confirmation of tumour-free margins) and can range between 0/2 to 2/2. The oncological validity rate will be defined as the percentage of patients who score 2/2 on the oncological validity scale.

SECONDARY OUTCOMES:
Process Feasibility will be determined by recruitment rate (The proportion of patients enrolled in the study versus the number eligible, up to n=30) | pre-operatively, an average of 2 years
Management Feasibility will be determined by the percentage of cases for which ICG was successfully obtained from pharmacy and prepared for the ENB-RIGGS procedure | pre-operatively, an average of 2 years
Resource Feasibility will be determined by the sum of the dollar costs of the ENB-RIGGS materials and personnel required to perform the procedure, divided by the number of participants. | pre-operatively, an average of 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Waël C. Hanna, MDCM, MBA, FRCSC, Principal Investigator — St. Joseph's Healthcare Hamilton / McMaster University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] National Lung Screening Trial Research Team; Aberle DR, Adams AM, Berg CD, Black WC, Clapp JD, Fagerstrom RM, Gareen IF, Gatsonis C, Marcus PM, Sicks JD. Reduced lung-cancer mortality with low-dose computed tomographic screening. N Engl J Med. 2011 Aug 4;365(5):395-409. doi: 10.1056/NEJMoa1102873. Epub 2011 Jun 29. PMID 21714641
- [Background] Finley RJ, Mayo JR, Grant K, Clifton JC, English J, Leo J, Lam S. Preoperative computed tomography-guided microcoil localization of small peripheral pulmonary nodules: a prospective randomized controlled trial. J Thorac Cardiovasc Surg. 2015 Jan;149(1):26-31. doi: 10.1016/j.jtcvs.2014.08.055. Epub 2014 Sep 16. PMID 25293355
- [Background] Hachey KJ, Colson YL. Current innovations in sentinel lymph node mapping for the staging and treatment of resectable lung cancer. Semin Thorac Cardiovasc Surg. 2014 Autumn;26(3):201-9. doi: 10.1053/j.semtcvs.2014.09.001. Epub 2014 Sep 16. PMID 25527014
- [Background] Okusanya OT, Holt D, Heitjan D, Deshpande C, Venegas O, Jiang J, Judy R, DeJesus E, Madajewski B, Oh K, Wang M, Albelda SM, Nie S, Singhal S. Intraoperative near-infrared imaging can identify pulmonary nodules. Ann Thorac Surg. 2014 Oct;98(4):1223-30. doi: 10.1016/j.athoracsur.2014.05.026. Epub 2014 Aug 5. PMID 25106680